CLINICAL TRIAL: NCT01310582
Title: Recovery Following Desflurane vs Sevoflurane for Outpatient Urologic Surgery in Elderly Females
Brief Title: Recovery Following Desflurane Versus Sevoflurane for Outpatient Urologic Surgery in Elderly Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hahnemann University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Michael Green, DO, Assistant Professor, Hahnemann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19326
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Ureteral Stent Occlusion; Exposure Laser; Ureterostomy; Functional Disturbance; Vaginal Diseases; Injury of Bladder; Excessive Repair; Calculi
Keywords: Sevoflurane; Desflurane
MeSH Terms: conditions — Vaginal Diseases; Calculi | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Active Comparator): During the surgery the subjects were given Desflurane, general anesthesia, that will keep the patient asleep during the surgery. The dosage form was inhalation gas, dosage equivalent to 1 MAC, frequency was once and the duration was throughout the surgery (30-45 minutes).
  Interventions: Drug: Desflurane
- Sevoflurane (Active Comparator): During the surgery the subjects were given Sevoflurane, general anesthesia, that will keep the patient asleep during the surgery. The dosage form was inhalation gas, dosage equivalent to 1 MAC, frequency was once and the duration was throughout the surgery (30-45 minutes).
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desflurane
  Arms: Desflurane
Drug: Sevoflurane
  Arms: Sevoflurane

SUMMARY:
Numerous studies demonstrate that patients have improved immediate recovery characteristics following desflurane anesthesia compared to other volatile agents, including sevoflurane. There is limited evidence in the literature to suggest that patients undergoing sevoflurane, compared to desflurane anesthesia, may suffer from limitation in function and cognitive ability for an undetermined, but prolonged period of time following surgery. These differences are not explained pharmacokinetically and may be a result of a direct neurotoxic effect of sevoflurane. An unresolved question is the time required for the ability to return to complex tasks, such as driving, following anesthesia. Commonly, patients are advised not to drive or make important decisions for 24 hours following anesthesia, but this is not well-studied and proscribed on an empiric, rather than scientific, basis with very limited data available.This study will better define recovery characteristics and characterize the severity and duration of cognitive impairment following sevoflurane or desflurane anesthesia after brief outpatient urologic surgery in elderly females using tests of cognitive ability coupled with performance on a driving simulator and cognitive task tests to objectively measure not only testing performance, but also cognitive effort in performing these tests.

DETAILED DESCRIPTION:
Following IRB-approved consent, 60 patients were be randomized (63 patients to be enrolled accounting for a <5% screen failure and <5% dropped patient rates) to receive either a desflurane or sevoflurane-based anesthetic for pelvic floor repair. The selection of the anesthetic gas (sevoflurane or desflurane) was determined by computer generated randomization. Only the Anesthesiologist or the CRNA knows which gas has been administered to the subject. All the investigators and the co-investigator who collected the research data were blinded to the gas selection.

Potential subjects were identified during the clinic visit in the Urology Department in Hahnemann University Hospital.

On the morning of the surgery, the study investigator who is a medical doctor asked the subjects to perform a baseline cognitive task tests to determine the baseline thinking process. The detailed description of the cognitive task is as following;

1. Mini-Mental Status Exam (MMSE): (10-15 minutes) This is a 30-item measure of global cognition (Folstein, Folstein & McHugh, 1975) that tests orientation to time and place, object naming, repetition, attention, recall, and following complex commands.
2. Trail Making Test Part A and Part B: Part A (3 minutes) of this measure (Army Individual Test Battery, 1944; Reitan & Wolfson, 1985) is a test of visual attention where the subjects must draw lines on a page connecting 25 consecutive number as quickly as possible. Part B (5 minutes) requires the subject to alternately sequence numbers and letters randomly distributed on a page into their ascending and alphabetical order as quickly as possible.
3. Digit Symbol Coding: (2 minutes) This subtest of the WAIS-III (Wechsler, 1997) consists of nine digit-symbol pairs followed by a list of digits. Under each digit the subject must write down the corresponding symbol as quickly as possible.
4. Hopkins Verbal Learning Test-Revised (HVLT-R): (8 minutes) Memory for verbal information will be assessed with this list learning task assessing immediate and delayed recall.
5. Stroop Color and Word Test: (5 minutes) This test (Stroop, 1935; Golden, 2002) measures cognitive control by asking subjects to suppress a habitual response in favor of an alternate response. Participants are shown a word and asked to name the color in which the word is written Total time expected for cognitive task tests is 28-33 min. If the patients' were able to drive and have been driving for at least one year, they were required to perform driving simulation. After performing the baseline cognitive task tests, baseline driving simulation (15 minutes) on the driving simulator.

After the baseline Cognitive Task Test and Virtual Driving Training session, the subjects underwent their planned surgery. The selection of the anesthetic gas was determined by a computer generated randomization list. The anesthesiologist or the CRNA in charge of the subject administered anesthesia. The investigators and the subjects were blinded to the anesthetic gas given. At the conclusion of the surgery, the anesthetic gas was shut down and the co-investigator was called into the OR to document the time the subjects take to open their eyes after the cessation of the gas.

At 30 minutes after discontinuation of the anesthetic gas, the subjects were asked to repeat the same sets of cognitive task tests (28-33 min).

And, at 2 hours after the surgery, the subjects repeated the cognitive tasks test (28-33 min) and the driving simulation (20 min) for patients who were able to drive.

On the next day of the surgery, the co-investigator had a telephone conversation with the subjects who were discharged home after the surgery. Modified Telephone Interview for Cognitive Status (TICS-M) was used to collect data (10 minutes). This is a 13-item telephone interview (Welsh, Breitner, & Magruder-Habib, 1993) for late-life cognitive assessment that includes tests of orientation, attention, working memory, praxis, sentence repetition, naming to verbal description, recent memory, word opposites, and an additional immediate and delayed recall of a 10-word list. The subjects' participation in the study ended after this follow-up telephone call.

The participants were followed for the duration up to 28 hours. The follow-up and participation in this study ended after 24-28 hours.

From date of randomization until the date of first documented progression, end of participation or date of death from any cause, whichever came first, assessed up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old, female subjects
* Scheduled for brief urologic surgery (Cyctoscopy, Ureteral stent, Laserlithotripsy, Ureteroscopy, Vaginal sling, Bladder injury repair, Rectocele repair and Stone extraction)
* Ability to read, write and speak English language
* Driving at least one year

Exclusion Criteria:

* Preexisting neurological impairment in thinking process
* Renal insufficiency or failure
* Lack of command of English language
* Inability to drive
* Motion Sickness

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Mychaskiw, DO, Principal Investigator — Professor and Chair, Department of Anesthesiology
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recuitment was done from May 2011 to May 2013 at the Drexel University College of Medicine/Hahnemann University Hospital, there is a subspecialty practice of urologic surgery and pelvic floor repairs in elderly females.
Pre-assignment Details: Participant enrollment performed during the subject's pre admission testing at Hahnemann Hospital. Consented subjects were approched again on the morning of their surgery and group assignment was done. No other events prior to randomization, which was determined by computer generated randomization.
Groups:
- Desflurane: During the surgery the subjects will be given Desflurane, general anesthesia, that will keep the patient asleep during the surgery. The dosage form is inhalation gas, dosage equivalent to 1 MAC, frequency is once and the duration is throughout the surgery (30-45 minutes).
- Sevoflurane: During the surgery the subjects will be given Sevoflurane, general anesthesia, that will keep the patient asleep during the surgery. The dosage form is inhalation gas, dosage equivalent to 1 MAC, frequency is once and the duration is throughout the surgery (30-45 minutes).
Period: Overall Study
Arm/Group | Desflurane | Sevoflurane
Started | 31 | 26
Completed | 31 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Six patients dropped out due to physician decision.
Groups:
- Total: Total of all reporting groups
Arm/Group | Desflurane | Sevoflurane | Total
Number analyzed (Participants) | 31 | 26 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 31 | 26 | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 68.2 (6.43) | 67.1 (6.11) | 67.6 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 26 | 57

OUTCOME MEASURES:

1. Primary Outcome: Time to Opening of Eyes
Time Frame: At 30-45 minutes, following discontinuation of volatile anesthetic at the end of surgery
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 31 | 26
seconds | 391.2 (250.04) | 446.5 (228.19)

2. Secondary Outcome: Time to Discharge From PACU
Time Frame: At 30-45 minutes, following discontinuation of volatile anesthetic at the end of surgery and transfer to PACU
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 31 | 26
Minutes | 95.0 (34.24) | 104.9 (49.82)

ADVERSE EVENTS:
Arm/Group | Desflurane | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/26
Other Adverse Events (participants affected / at risk) | 0/31 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No